CLINICAL TRIAL: NCT01250145
Title: A Multiple-Dose Study to Evaluate Skin Irritation and Sensitization of Teriparatide Administered Transdermally in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13764; I2Y-EW-GHFO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY333334 + placebo (Experimental): Part A:
  Both a placebo and an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days
  Part B:
  Induction phase: Both a placebo and an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks
  Rest phase: 2 weeks with no patch application
  Challenge phase: 80 microgram active patch given once for at least 6 hours
  Interventions: Drug: LY333334; Drug: Placebo

INTERVENTIONS:
Drug: LY333334 — Transdermal patch
Drug: Placebo — Transdermal patch

SUMMARY:
This study is a Phase 1, multi-center, 2-part, subject- and investigator-blind, randomized, placebo-controlled, multiple dose study of transdermal teriparatide (80-µg dose) in healthy postmenopausal women. Part A will examine the cumulative irritation and adherence of the transdermal patch, and Part B will examine skin sensitization and adherence. Two separate groups of subjects will be enrolled for Part A and Part B of the study. All screening procedures will take place up to 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy postmenopausal females, as determined by medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests (for example, subjects who have osteoporosis or stable and/or controlled hyperlipidemia, hypertension, and/or hypothyroidism may be entered if that investigator judges it appropriate for participation in this study).
* Postmenopausal women include women with at least 6-weeks postsurgical bilateral oophorectomy with or without hysterectomy, confirmed by medical history, or spontaneous amenorrhea for at least 6 to 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (eg, oral contraceptives, hormones, gonadotropin-releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy) and a follicle-stimulating hormone level greater than 40 mIU/mL.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have a sitting blood pressure and pulse rate that are judged to be not clinically significant by the investigator.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Eli Lilly and Company (Lilly) and the ethical review board (ERB) governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 3 months from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known hypersensitivity to teriparatide or to any of its excipients.
* Are persons who have previously completed or withdrawn from this study or any other study investigating teriparatide patch.
* Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Have a history of breast cancer within the past 10 years or other types of carcinoma within the past 5 years, except for excised superficial skin tumors and adequately treated in situ carcinoma of cervix.
* Have an average weekly alcohol intake that exceeds 14 units per week,

  (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Have hyperparathyroidism or hypoparathyroidism.
* Have hyperthyroidism.
* Have hypercalciuria (24-hour collection above 300 mg/day).
* Have hypercalcemia (above the upper limit of reference range).
* Have a history of bone diseases such as Paget's disease of bone, bone carcinoma, bone metastases, metabolic bone disease other than osteoporosis, or unexplained elevation in serum alkaline phosphatase level.
* Have a history of external beam or implant radiation involving the skeleton.
* Have a history of recurrent nephrolithiasis, or a single episode within the past 5 years. Eligible subjects who have had an episode within the past 5 to 10 years must have a kidney-ureter-bladder X-ray of the abdominal area within 1 month prior to enrollment in the study, which indicates no existing stone.
* Have a history of bleeding disorder within the past 3 years.
* Are currently using therapies for osteoporosis; or using hormone replacement therapy or bisphosphonates during the previous 3 months. Women receiving short-term hormone therapy for the treatment of moderate to severe menopausal symptoms may be enrolled if their postmenopausal status is confirmed by inclusion criterion.
* Have presence of a dermatologic disease that might interfere with the evaluation of the test site reaction; and clinically significant scars, wounds, or discoloration, or abnormalities of the skin at or near the intended site of electrode application (for example, porphyria, atopy, psoriasis, vitiligo).
* Have a history of severe skin infection within the past year in the opinion of the investigator.
* Have a history of skin allergy or hypersensitivity to tapes or adhesives, in the opinion of the investigator.
* Have a history of significant dermatologic cancers (for example, melanoma, squamous cell carcinoma), except basal-cell carcinomas that were superficial and did not involve the investigative site.
* Have an obvious difference in skin color between arms or the presence of a skin condition, excessive hair at the application sites, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug.
* Have implanted or externally mounted electrical or electronic medical devices (for example, pacemakers).
* Have used topical analgesics or topical corticosteroids within 3 weeks of study enrollment.
* Have taken antihistamines within 72 hours prior to dosing.
* Any other condition which, in the opinion of the investigator, would preclude participation in the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schenefeld
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devon, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- LY333334 + Placebo: Part A: Part A:
  Both a placebo and an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days
- LY333334 + Placebo: Part B: Part B:
  Induction phase: Both a placebo and an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks
  Rest phase: 2 weeks with no patch application
  Challenge phase: 80 microgram active patch given once for at least 6 hours
Period: Overall Study
Arm/Group | LY333334 + Placebo: Part A | LY333334 + Placebo: Part B
Started | 41 | 210
Completed | 39 | 205
Not Completed | 2 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY333334 + Placebo: Part A | LY333334 + Placebo: Part B | Total
Number analyzed (Participants) | 41 | 210 | 251
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.1) | 59.9 (6.7) | 59.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 210 | 251
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 38 | 201 | 239
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 33 | 74
  Germany | 0 | 103 | 103
  United Kingdom | 0 | 74 | 74

OUTCOME MEASURES:

1. Primary Outcome: Part A - Cumulative Skin Irritation by Draize Score
Description: Number of evaluation points (patches) showing defined Draize score. Erythema and edema were used to determine skin irritation. Score 0 = No Erythema/Edema; Score 1 = Very slight Erythema/Edema (barely perceptible); Score 2 = Well defined Erythema/Edema (edges of area well defined by definite raising); Score 3 = Moderate to Severe Erythema/Edema (raised approximately 1 millimeter [mm]).
Time Frame: Day 1 through Day 22
Population: All participants who entered the study and received patches are included in the analysis.
Measure: Number; unit: patches with Draize scores
Units Other Than Participants: Patches
Groups:
- Part A: Active Patch - Prior to Patch Application: Part A: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores prior to patch application.
- Part A: Active Patch - 1 Hour Post Patch Removal: Part A: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores 1 hour after patch removal.
- Part A: Active Patch - 24 Hours Post Patch Application: Part A: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores 24 hours after patch application.
- Part A: Placebo Patch - Prior to Patch Application: Part A: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores prior to patch application.
- Part A: Placebo Patch - 1 Hour Post Patch Removal: Part A: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores 1 hour after patch removal.
- Part A: Placebo Patch - 24 Hours Post Patch Application: Part A: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days. Scores 24 hours after patch application.
Arm/Group | Part A: Active Patch - Prior to Patch Application | Part A: Active Patch - 1 Hour Post Patch Removal | Part A: Active Patch - 24 Hours Post Patch Application | Part A: Placebo Patch - Prior to Patch Application | Part A: Placebo Patch - 1 Hour Post Patch Removal | Part A: Placebo Patch - 24 Hours Post Patch Application
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41 | 41
Number analyzed (Patches) | 888 | 890 | 887 | 888 | 890 | 887
patches with Draize scores
  Erythema: Score 0 | 299 | 40 | 146 | 390 | 69 | 205
  Erythema: Score 1 | 523 | 674 | 633 | 452 | 713 | 601
  Erythema: Score 2 | 65 | 176 | 106 | 45 | 108 | 79
  Erythema: Score 3 | 1 | 0 | 2 | 1 | 0 | 2
  Edema: Score 0 | 604 | 113 | 370 | 716 | 298 | 539
  Edema: Score 1 | 270 | 600 | 454 | 166 | 511 | 322
  Edema: Score 2 | 13 | 175 | 62 | 5 | 80 | 26
  Edema: Score 3 | 1 | 1 | 1 | 1 | 0 | 0

2. Secondary Outcome: Part A - Patch Adhesion Score
Description: Number of patches with adhesion score. Score 0 = ≥90% adhered (essentially no lift off the skin); Score 1= ≥75% to <90% adhered (some edges only lifting off the skin); Score 2 = ≥50% to <75% adhered (less than half of the patch lifting off the skin); Score 3 = >0% to <50% adhered but not detached (more than half of the patch lifting off the skin without falling off); Score 4 = 0% adhered - patch detached (patch completely off the skin).
Time Frame: Day 1 through Day 22
Population: All randomized participants who received a patch.
Measure: Number; unit: patches with adhesive score
Units Other Than Participants: Patches
Groups:
- Active Patch: Part A: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days
- Placebo Patch: Part A: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, for 22 days
Arm/Group | Active Patch | Placebo Patch
Number analyzed (Participants) | 41 | 41
Number analyzed (Patches) | 889 | 889
patches with adhesive score
  Score 0 | 879 | 882
  Score 1 | 8 | 7
  Score 2 | 1 | 0
  Score 3 | 0 | 0
  Score 4 | 1 | 0

3. Primary Outcome: Part B - Skin Irritation and Sensitization by Draize Score
Description: Number of evaluation points (patches) showing defined Draize score. Erythema and edema were used to determine skin irritation and sensitization. Score 0 = No Erythema/Edema; Score 1 = Very slight Erythema/Edema (barely perceptible); Score 2 = Well defined Erythema/Edema (edges of area well defined by definite raising); Score 3 = Moderate to Severe Erythema/Edema (raised approximately 1 mm); Score 4 = Severe Edema (raised more than 1 mm and extending beyond area of exposure).
Time Frame: Days 1 - 19 and 34 - 37
Population: All participants who entered the study and received patches are included in the analysis.
Measure: Number; unit: patches with Draize scores
Units Other Than Participants: Patches
Groups:
- Part B: Active Patch - Prior to Patch Application: Part B: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores prior to patch application.
- Part B: Active Patch - 1 Hour Post Patch Removal: Part B: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores 1 hour after patch removal.
- Part B: Active Patch - 24 Hours Post Patch Application: Part B: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores 24 hours after patch application.
- Part B: Placebo Patch - Prior to Patch Application: Part B: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores prior to patch application.
- Part B: Placebo Patch - 1 Hour Post Patch Removal: Part B: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores 1 hour after patch removal.
- Part B: Placebo Patch - 24 Hours Post Patch Application: Part B: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks. Scores 24 hours after patch application.
Arm/Group | Part B: Active Patch - Prior to Patch Application | Part B: Active Patch - 1 Hour Post Patch Removal | Part B: Active Patch - 24 Hours Post Patch Application | Part B: Placebo Patch - Prior to Patch Application | Part B: Placebo Patch - 1 Hour Post Patch Removal | Part B: Placebo Patch - 24 Hours Post Patch Application
Number analyzed (Participants) | 210 | 210 | 210 | 210 | 210 | 210
Number analyzed (Patches) | 2479 | 2479 | 2474 | 2474 | 2474 | 2469
patches with Draize scores
  Erythema: Score 0 | 1399 | 122 | 436 | 1525 | 271 | 784
  Erythema: Score 1 | 1050 | 1503 | 1899 | 924 | 1698 | 1578
  Erythema: Score 2 | 30 | 840 | 138 | 25 | 495 | 107
  Erythema: Score 3 | 0 | 14 | 1 | 0 | 10 | 0
  Edema: Score 0 | 2280 | 930 | 1759 | 2330 | 1572 | 2014
  Edema: Score 1 | 197 | 1141 | 661 | 143 | 766 | 435
  Edema: Score 2 | 2 | 399 | 53 | 1 | 136 | 19
  Edema: Score 3 | 0 | 5 | 1 | 0 | 0 | 1
  Edema: Score 4 | 0 | 4 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part B - Patch Adhesion Score
Description: as for outcome 2
Time Frame: Days 1 - 19 and 34 - 37
Population: All randomized participants who received a patch.
Measure: Number; unit: patches with adhesive score
Units Other Than Participants: Patches
Groups:
- Active Patch: Part B: an 80 microgram active patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks.
  Rest phase: 2 weeks with no patch application
  Challenge phase: 80 microgram active patch given once for at least 6 hours
- Placebo Patch: Part B: a placebo patch will be applied to the same arm for at least 6 hours daily, test arms will be alternated daily, 4 times a week for 3 weeks.
  Rest phase: 2 weeks with no patch application
  Challenge phase: placebo patch given once for at least 6 hours
Arm/Group | Active Patch | Placebo Patch
Number analyzed (Participants) | 210 | 210
Number analyzed (Patches) | 2683 | 2678
patches with adhesive score
  Score 0 | 2608 | 2608
  Score 1 | 40 | 31
  Score 2 | 13 | 17
  Score 3 | 9 | 17
  Score 4 | 13 | 5

ADVERSE EVENTS:
Arm/Group | LY333334 + Placebo: Part A | LY333334 + Placebo: Part B
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/210
Other Adverse Events (participants affected / at risk) | 31/41 | 157/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY333334 + Placebo: Part A (N=41) | LY333334 + Placebo: Part B (N=210)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY333334 + Placebo: Part A (N=41) | LY333334 + Placebo: Part B (N=210)
Nausea (Gastrointestinal disorders) | 0 (0) | 17 (18)
Application site erythema (General disorders) | 0 (0) | 31 (79)
Application site pain (General disorders) | 4 (6) | 12 (19)
Application site pruritus (General disorders) | 11 (25) | 33 (88)
Fatigue (General disorders) | 0 (0) | 13 (13)
Nasopharyngitis (Infections and infestations) | 0 (0) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 12 (14)
Headache (Nervous system disorders) | 5 (9) | 53 (74)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 13 (17)
Constipation (Gastrointestinal disorders) | 8 (9) | 0 (0)
Application site erosion (General disorders) | 8 (11) | 0 (0)
Application site vesicles (General disorders) | 3 (4) | 0 (0)
Nasal congestion (General disorders) | 3 (3) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days